CLINICAL TRIAL: NCT00981877
Title: Probiotics in the Management of Acute Rotavirus Diarrhea in Bolivian Children: Randomized Double-blind, Controlled Trial Using Two Different Preparations
Brief Title: Probiotics in the Management of Acute Rotavirus Diarrhea in Bolivian Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Pediatrico Albina de Patino (Other)
Collaborators: Instituto de Nutrición y Tecnología de los Alimentos (Other)
Responsible Party: Giuseppe Grandy Aranda, Centro Pediatrico Albina de Patino/ Departamento de Gastroenterologia y Nutricion
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: protrota2007
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Diarrhea; Rotavirus Infection
Keywords: acute diarrhea; rotavirus; probiotic; children
MeSH Terms: conditions — Diarrhea; Rotavirus Infections

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): This group will receive S. Boulardii Probiotic and Oral rehydration as needed
  Interventions: Drug: GB (Florestor)
- 2 (Active Comparator): This group will receive a mixed Probiotic preparation and oral rehydration as needed
  Interventions: Drug: GRALB
- 3 (Placebo Comparator): This group will receive a placebo, and oral rehydration as needed
  Interventions: Drug: GC (placebo)

INTERVENTIONS:
Drug: GB (Florestor) — S. Boulardii preparation of 1 gram twice daily for 5 days
  Other Names: Florestor, Bioflora
  Arms: 1
Drug: GRALB — mixed probiotic preparation 1 gram twice daily for 5 days.
  Other Names: Probiotik, mixed probiotic
  Arms: 2
Drug: GC (placebo) — Placebo 1 gram twice daily for 5 days.
  Other Names: Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to determine the effect of probiotics in rotavirus acute diarrhea in children. The investigators will compare the effect of two different probiotics products.

DETAILED DESCRIPTION:
Acute diarrhea remains being the second most frequent infectious condition in children, producing a high number of admissions yearly. In children below one year of age, rotavirus represents the main etiologic agent, both in developed and developing countries. In Bolivia, acute diarrhea affects about 30% of the group below 5 years of age. Probiotics appear as one of the alternatives currently under discussion. Also, evidence available suggests that probiotics shorten the time of diarrhea and therefore the time of rotavirus excretion. In daily practice, we are often limited by the type and number of probiotics products locally available; moreover, information about combined products is scarce. With this in mind, in this study we compared the efficacy of two commercially available products.

ELIGIBILITY:
Inclusion Criteria:

* Positive stool sample for rotavirus test

Exclusion Criteria:

* Severe malnourishment
* Severe dehydration
* Use of antibiotics, probiotics or nitazoxanide 2 weeks before admission
* Systemic infections
* Severe chronic disease
* Mixed enteric infections besides rotavirus

Ages: 1 Month to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | within the first 72 hours during hospitalization

SECONDARY OUTCOMES:
Duration of fever | the first 72 hours during hospitalization
Duration of vomiting | the first 72 hours during hospitalization
Duration of hospitalization | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Soria, MD, Study Director — Centro Pediatrico Albina Patino; Giuseppe E Grandy, Md, Principal Investigator — Centro Pediatrico Albina Patino - Instituto de Nutricion y Tecnologia de los Alimentos
Locations (1):
- Centro Pediatrico Albina Patino, Cochabamba, Departamento de Cochabamba, Bolivia

REFERENCES:
- [Derived] Smithline HA, Donnino M, Greenblatt DJ. Pharmacokinetics of high-dose oral thiamine hydrochloride in healthy subjects. BMC Clin Pharmacol. 2012 Feb 4;12:4. doi: 10.1186/1472-6904-12-4. PMID 22305197
- [Derived] Waldvogel S, Pedrazzini B, Vaucher P, Bize R, Cornuz J, Tissot JD, Favrat B. Clinical evaluation of iron treatment efficiency among non-anemic but iron-deficient female blood donors: a randomized controlled trial. BMC Med. 2012 Jan 24;10:8. doi: 10.1186/1741-7015-10-8. PMID 22272750
- [Derived] Savolainen-Kopra C, Haapakoski J, Peltola PA, Ziegler T, Korpela T, Anttila P, Amiryousefi A, Huovinen P, Huvinen M, Noronen H, Riikkala P, Roivainen M, Ruutu P, Teirila J, Vartiainen E, Hovi T. Hand washing with soap and water together with behavioural recommendations prevents infections in common work environment: an open cluster-randomized trial. Trials. 2012 Jan 16;13:10. doi: 10.1186/1745-6215-13-10. PMID 22243622
- [Derived] Wiseman V, Mangham LJ, Cundill B, Achonduh OA, Nji AM, Njei AN, Chandler C, Mbacham WF. A cost-effectiveness analysis of provider interventions to improve health worker practice in providing treatment for uncomplicated malaria in Cameroon: a study protocol for a randomized controlled trial. Trials. 2012 Jan 6;13:4. doi: 10.1186/1745-6215-13-4. PMID 22225699
- [Derived] Husebye EE, Lyberg T, Opdahl H, Aspelin T, Stoen RO, Madsen JE, Roise O. Intramedullary nailing of femoral shaft fractures in polytraumatized patients. a longitudinal, prospective and observational study of the procedure-related impact on cardiopulmonary- and inflammatory responses. Scand J Trauma Resusc Emerg Med. 2012 Jan 5;20:2. doi: 10.1186/1757-7241-20-2. PMID 22221511
- [Derived] Pontes-Arruda A, Martins LF, de Lima SM, Isola AM, Toledo D, Rezende E, Maia M, Magnan GB; Investigating Nutritional Therapy with EPA, GLA and Antioxidants Role in Sepsis Treatment (INTERSEPT) Study Group. Enteral nutrition with eicosapentaenoic acid, gamma-linolenic acid and antioxidants in the early treatment of sepsis: results from a multicenter, prospective, randomized, double-blinded, controlled study: the INTERSEPT study. Crit Care. 2011 Jun 9;15(3):R144. doi: 10.1186/cc10267. PMID 21658240
- [Derived] Grandy G, Medina M, Soria R, Teran CG, Araya M. Probiotics in the treatment of acute rotavirus diarrhoea. A randomized, double-blind, controlled trial using two different probiotic preparations in Bolivian children. BMC Infect Dis. 2010 Aug 25;10:253. doi: 10.1186/1471-2334-10-253. PMID 20735858